CLINICAL TRIAL: NCT04541108
Title: A Phase 0 Master Protocol Using the CIVO® Platform to Evaluate Intratumoral Microdoses of Anti-Cancer Therapies in Patients With Solid Tumors
Brief Title: Phase 0 Master Protocol for CIVO Intratumoral Microdosing of Anti-Cancer Therapies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Presage Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBI-MST-01; MST01-TAK-02 (NCT06062602) (Other: Presage Biosciences); MST01-MSD-03 (Other: Presage Biosciences); MST01-AZN-05 (NCT06366451) (Other: Presage Biosciences)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor
Keywords: HNSCC; SCCHN; lymphoma; sarcoma; breast adenocarcinoma; melanoma; intratumoral microdosing; microdose injection; microdosing; in vivo oncology; in vivo drug sensitivity; tumor microenvironment; multiplexed immunohistochemistry; head and neck cancer; pharmacodynamic biomarkers; CIVO; master protocol; precision oncology; soft tissue sarcoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoma; Sarcoma; Melanoma; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This Master Protocol is designed as an umbrella concept trial for the ongoing evaluation of multiple agents in individual CIVO Phase 0 substudies. Based on regulatory guidance on Phase 0 clinical trial design, approximately up to 15 participants are planned to be enrolled in each substudy in order to complete with approximately up to 12 evaluable tumor samples. Each substudy is considered an "Experimental Arm" with specified tumor types, inclusion and exclusion criteria, and investigational agents and combinations to be evaluated. Tumor type examples accessible for CIVO injection include, but may not be limited to, Head and Neck Cancer, Melanoma, Soft Tissue Sarcoma, Breast Cancer, or Lymphoma. Comparisons will not be made between experimental arms/substudies.
  The following substudy(ies) is(are) currently active:
  - MST01-AZN-05 (NCT06366451) evaluating rilvegostomig, volrustomig, sabestomig, and pembrolizumab.
  New substudies will be continuously added as they become active.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rilvegostomig, Volrustomig, Sabestomig, Pembrolizumab (Experimental): HNSCC patients presenting with a surface accessible lesion who are scheduled for tumor and/or regional node dissection as part of their standard treatment will be injected one to three days prior to surgery using the CIVO device. The planned injection scheme includes: vehicle control and microdoses of rilvegostomig, volrustomig, sabestomig, and pembrolizumab alone.
  Interventions: Biological: Rilvegostomig; Biological: Volrustomig; Biological: Sabestomig; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Rilvegostomig — Intratumoral microdose injection by the CIVO device.
  Other Names: AZD2936
Biological: Volrustomig — Intratumoral microdose injection by the CIVO device.
  Other Names: MEDI5752
Biological: Sabestomig — Intratumoral microdose injection by the CIVO device.
  Other Names: AZD7789
Biological: Pembrolizumab — Intratumoral microdose injection by the CIVO device.
  Other Names: Keytruda, MK-3475

SUMMARY:
This is a multi-center, open-label Phase 0 Master Protocol designed to study the localized pharmacodynamics (PD) of anti-cancer therapies within the tumor microenvironment (TME) when administered intratumorally in microdose quantities via the CIVO device in patients with surface accessible solid tumors for which there is a scheduled surgical intervention. CIVO stands for Comparative In Vivo Oncology. Multiple substudies will include specified investigational agents and combinations to be evaluated.

DETAILED DESCRIPTION:
CIVO is a research tool composed of a hand-held single-use sterile injector coupled with fluorescent tracking microspheres called CIVO GLO that mark the sites of drug microdose injection, enabling rapid assessment of multiple oncology drugs or drug combinations simultaneously within a patient's tumor. Tumor responses to cancer treatments are highly context-specific and often involve complex interactions between the anti-cancer therapy, genetically diverse tumor cells, and a heterogeneous TME. This complexity is rarely modeled accurately in preclinical translational models of cancer. By utilizing intratumoral microdose injections with CIVO in advance of scheduled surgical intervention, this study will evaluate anti-cancer therapies directly in patients each with their own unique tumor genomic profile, intact TME, and immune system functional status. Because the platform delivers microdose amounts of each test agent or combination directly into the patient's tumor tissue, hypotheses can be tested earlier in the drug development process, consistent with the goals of the 2006 FDA Exploratory IND Guidance for Industry.

The CIVO device penetrates solid tumors and simultaneously delivers subtherapeutic microdoses of up to eight anti-cancer agents or combinations of anti-cancer agents co-injected with CIVO GLO into discrete regions of the tumor as drug columns. At the time of the planned surgical intervention (at least four hours to up to seven days after the CIVO microdose injection), the injected tumor tissue is then excised and tumor responses are assessed via histological staining of tumor cross-sections sampled perpendicular to each injection column. Co-injection with CIVO GLO enables identification of each injection site during resection as well as in tissues stained for analysis. This Phase 0 Master Protocol is aimed at distinguishing promising candidates earlier in the drug development process while also avoiding systemic toxicities associated with typical clinical exposures to these therapies.

ELIGIBILITY:
*This list is representative of study inclusion/exclusion criteria. Each substudy may include variations on these criteria.

Inclusion Criteria:

1. Ability and willingness to comply with the study's visit and assessment schedule.
2. Male or female ≥ 18 years of age at Visit 1 (Screening).
3. Pathologic diagnosis of [solid tumors] indicated in the relevant substudy(ies).
4. Ability and willingness to provide written informed consent. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
5. At least one lesion (primary tumor, recurrent tumor, or metastatic lymph node) that is surface accessible for CIVO injection that contains viable minimum tumor tissue volume and characteristics (e.g., based on clinical evaluation, available pre-operative imaging, pre-injection ultrasound imaging, or pathology reports indicating lesion with appropriate viable tumor volume without excessive cysts or necrosis) and for which there is a planned surgical intervention. The patient's presentation, surgical and pathology plan may determine whether a lesion is eligible with respect to a given CIVO MID needle configuration.
6. Female patients who:

   * Are postmenopausal for at least one year before the screening visit, OR
   * Are surgically sterile, OR
   * Are of childbearing potential who agree to practice a highly effective method of contraception from the time of signing the Informed Consent Form (ICF) and during study participation OR agree to completely abstain from heterosexual intercourse.
   * Agree to refrain from donating ova during study participation.

Male patients, even if surgically sterile (i.e., status post-vasectomy), who:

* Agree to practice effective barrier contraception from the time of signing the ICF and during study participation OR agree to completely abstain from heterosexual intercourse.
* Agree to refrain from donating sperm during study participation.

Exclusion Criteria:

1. Tumors near or involving critical structures for which, in the opinion of the treating clinician, injection would pose undue risk to the patient.
2. Female patients who are:

   * Both lactating and breastfeeding, OR
   * Have a positive β-subunit human chorionic gonadotropin (β-hCG) pregnancy test at screening verified by the Investigator.
3. Any uncontrolled intercurrent illness, condition, serious medical or psychiatric illness, or circumstance that, in the opinion of the Investigator, could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of Selected Pharmacodynamic Biomarkers as Specified in Substudies by IHC, ISH, and/or Spatial Biology Platforms | 4 hours-7 days after microdose injection
  Quantification of biomarker-positive and biomarker-negative cells will be performed within the tumor microenvironment around each of the injection sites in each resected patient sample by IHC, ISH, or spatial biology platforms. An aggregate analysis of this quantification may be done across patient samples in each substudy to evaluate trends in tumor response. The biomarkers evaluated may include, but are not limited to biomarkers for cell death (e.g. cleaved caspase 3), T-cells (e.g. CD3, CD8/Granzyme B, CD4), natural killer (NK)/myeloid cells (e.g. CD56/Granzyme B, CD86, CD68, CD163), and proinflammatory cytokines (e.g., interferon gamma, tumor necrosis factor alpha, interferon gamma-induced protein 10).

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | Up to 28 days after microdose injection
  Relationship of AE to study drug(s) or CIVO device will be determined using an AE Relatedness Grading System.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Presage Biosciences
Locations (12):
- United States (12):
  - UC Davis, Sacramento, California
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - LSU Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - UC Health, Cincinnati, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Charleston, South Carolina
  - UT Health, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derry JMJ, Burns C, Frazier JP, Beirne E, Grenley M, DuFort CC, Killingbeck E, Leon M, Williams C, Gregory M, Houlton J, Clayburgh D, Swiecicki P, Huszar D, Berger A, Klinghoffer RA. Trackable Intratumor Microdosing and Spatial Profiling Provide Early Insights into Activity of Investigational Agents in the Intact Tumor Microenvironment. Clin Cancer Res. 2023 Sep 15;29(18):3813-3825. doi: 10.1158/1078-0432.CCR-23-0827. PMID 37389981
- [Background] Gundle KR, Deutsch GB, Goodman HJ, Pollack SM, Thompson MJ, Davis JL, Lee MY, Ramirez DC, Kerwin W, Bertout JA, Grenley MO, Sottero KHW, Beirne E, Frazier J, Dey J, Ellison M, Klinghoffer RA, Maki RG. Multiplexed Evaluation of Microdosed Antineoplastic Agents In Situ in the Tumor Microenvironment of Patients with Soft Tissue Sarcoma. Clin Cancer Res. 2020 Aug 1;26(15):3958-3968. doi: 10.1158/1078-0432.CCR-20-0614. Epub 2020 Apr 16. PMID 32299817
- [Background] Klinghoffer RA, Bahrami SB, Hatton BA, Frazier JP, Moreno-Gonzalez A, Strand AD, Kerwin WS, Casalini JR, Thirstrup DJ, You S, Morris SM, Watts KL, Veiseh M, Grenley MO, Tretyak I, Dey J, Carleton M, Beirne E, Pedro KD, Ditzler SH, Girard EJ, Deckwerth TL, Bertout JA, Meleo KA, Filvaroff EH, Chopra R, Press OW, Olson JM. A technology platform to assess multiple cancer agents simultaneously within a patient's tumor. Sci Transl Med. 2015 Apr 22;7(284):284ra58. doi: 10.1126/scitranslmed.aaa7489. PMID 25904742
- [Background] Frazier JP, Bertout JA, Kerwin WS, Moreno-Gonzalez A, Casalini JR, Grenley MO, Beirne E, Watts KL, Keener A, Thirstrup DJ, Tretyak I, Ditzler SH, Tripp CD, Choy K, Gillings S, Breit MN, Meleo KA, Rizzo V, Herrera CL, Perry JA, Amaravadi RK, Olson JM, Klinghoffer RA. Multidrug Analyses in Patients Distinguish Efficacious Cancer Agents Based on Both Tumor Cell Killing and Immunomodulation. Cancer Res. 2017 Jun 1;77(11):2869-2880. doi: 10.1158/0008-5472.CAN-17-0084. Epub 2017 Mar 31. PMID 28364003
- [Background] Dey J, Kerwin WS, Grenley MO, Casalini JR, Tretyak I, Ditzler SH, Thirstrup DJ, Frazier JP, Pierce DW, Carleton M, Klinghoffer RA. A Platform for Rapid, Quantitative Assessment of Multiple Drug Combinations Simultaneously in Solid Tumors In Vivo. PLoS One. 2016 Jun 30;11(6):e0158617. doi: 10.1371/journal.pone.0158617. eCollection 2016. PMID 27359113
- [Background] Moreno-Gonzalez A, Olson JM, Klinghoffer RA. Predicting responses to chemotherapy in the context that matters - the patient. Mol Cell Oncol. 2015 Jun 10;3(1):e1057315. doi: 10.1080/23723556.2015.1057315. eCollection 2016 Jan. PMID 27308571
- [Derived] Carideo Cunniff E, Sato Y, Mai D, Appleman VA, Iwasaki S, Kolev V, Matsuda A, Shi J, Mochizuki M, Yoshikawa M, Huang J, Shen L, Haridas S, Shinde V, Gemski C, Roberts ER, Ghasemi O, Bazzazi H, Menon S, Traore T, Shi P, Thelen TD, Conlon J, Abu-Yousif AO, Arendt C, Shaw MH, Okaniwa M. TAK-676: A Novel Stimulator of Interferon Genes (STING) Agonist Promoting Durable IFN-dependent Antitumor Immunity in Preclinical Studies. Cancer Res Commun. 2022 Jun 23;2(6):489-502. doi: 10.1158/2767-9764.CRC-21-0161. eCollection 2022 Jun. PMID 36923556